CLINICAL TRIAL: NCT03810547
Title: A Comparative Study Between Spinal and General Anesthesia for Abdominoplasty.
Brief Title: Abdominoplasty Under Spinal Anesthesia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Ayman Anis Metry, Assistant professor, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: ASUH1011/17
Record Dates: First submitted 2019-01-10; First posted 2019-01-18 (Actual); Last update posted 2019-01-22 (Actual); Status verified 2019-01

CONDITIONS: Spinal Anesthesia Suitability for Abdominoplasty
Keywords: Abdominoplasty; spinal anesthesia; general anesthesia; postoperative pain
MeSH Terms: conditions — Pain, Postoperative | interventions — Propofol; Ketamine

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Spinal anesthesia (Active Comparator): Patients undergoing abdominoplasty under spinal anesthesia may need to drug administration like propofol or ketamine or change anesthesia to general anesthesia.
  Interventions: Drug: Propofol 10 Mg/mL Intravenous Emulsion
- General anesthesia (No Intervention): General anesthesia for abdominoplasty

INTERVENTIONS:
Drug: Propofol 10 Mg/mL Intravenous Emulsion — when spinal anesthesia is not satisfactory intervention drugs are used
  Other Names: ketamine
  Arms: Spinal anesthesia

SUMMARY:
100 patients undergoing abdominoplasty under spinal anesthesia. 100 patients undergoing abdominoplasty under general anesthesia

DETAILED DESCRIPTION:
200 patients, American Society of Anesthesiologists (ASA) physical status classes I and II, were enrolled in this feasible study. All patients were subjected to abdominoplasty operation under spinal anesthesia or general anesthesia. Any intraoperative complications like hypotension, bradycardia, pain, nausea and vomiting related to spinal anesthesia were managed and recorded. Postoperative visual analogue scale (VAS) was used to assess pain severity and the need for analgesia to be administered.

ELIGIBILITY:
Inclusion Criteria:

* All patients between 18-55 years
* ASA I and II

Exclusion Criteria:

* BMI more than 35 years
* Contraindications for regional anesthesia

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 200 (Actual)
Dates: Start 2017-01-30 (Actual); Primary Completion 2018-04-30 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
Change in Pain sensation: Visual analogue scale | pain assessment during the operation and every 4 hours for 12 hours
  Visual analogue scale for Pain assessment from 1 with least pain to 10 with maximum pain felt
Patients satisfaction: Satisfaction score changes | Intraoperative assessment every 30 minutes till end of surgery.
  Satisfaction score with maximum score is fully satisfied and least is completely disagree

CONTACTS AND LOCATIONS:
Locations (1):
- Ain Shams University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No